CLINICAL TRIAL: NCT02392481
Title: An Exploratory, Prospective, Non-interventional Study Comparing Biomarker Signatures Between Patients With Asthma and Healthy Volunteers and to Investigate Biomarkers Associated With Known Phenotypes Across Asthma Severities
Brief Title: Asthma Biomarker Study
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 352.2087
Record Dates: First submitted 2015-03-18; First posted 2015-03-19 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2017-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and sputum

GROUPS / COHORTS (4):
- Healthy subjects
  Interventions: Procedure: Biofluid sampling
- Mild asthma
- Moderate asthma
- Severe asthma

INTERVENTIONS:
Procedure: Biofluid sampling
  Groups: Healthy subjects

SUMMARY:
The main objective of the trial is to explore if any of the biomarkers assessed are sensitively linked to the asthma phenotypes. This would potentially alone or in addition to other clinical or biofluid markers indicate if and how asthma endotypes are linked to phenotype such as eosinophilic, neutrophilic, or paucigranulocytic phenotypes. Further exploratory markers will be analysed for better understanding of physiological levels of proteins and markers playing a role in regard to disease characterization in asthma. As a basis for further development of a biomarker for asthma, The sponsor plans to conduct this exploratory biomarker trial to determine levels and reference ranges of biomarkers potentially associated with asthma phenotypes. The trial aims at generating a panel of serum biomarkers that can be evaluated in subsequent interventional studies. The longitudinal design will be used to ascertain stability and test-retest reliability.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

Body mass index (BMI) >=18 and <= 40 Non-smokers or ex-smokers with a cigarette smoking history of <= 10 pack years and smoking cessation for at least one year prior to enrolment Able to perform all trial related procedures including acceptable spirometry and production of induced sputum samples

Additional inclusion criteria for subject with asthma:

A minimum of one year history of asthma (physician diagnosed). Forced Expiratory Volume in one second (FEV1) reversibility of at least 12% above baseline at screening, unless documented in prior 12 months Methacholine response: concentration of <=8mg/ml to decrease FEV1 by 20% (PC20) at screening, unless documented in prior 12 months Stable asthma treatment for a period of 3 months (mild to moderate asthma) or 4 weeks (severe asthma).

Further Inclusion criteria apply.

Exclusion criteria:

Significant conditions or medical conditions that could influence the results of the study or the patient's ability to participate in the study Malignancy requiring resection, radiation or chemotherapy within 5 years prior to screening Planned surgery during the trial Blood donation of more than 400ml within 4 weeks of starting trial or during the trial Subjects unable or unwilling to comply with the medication, lifestyle or dietary requirements of the trial Pregnant or nursing women History of cystic fibrosis Clinically significant bronchiectasis Acute or chronic infections including hepatitis, HIV and tuberculosis Thoracotomy with pulmonary resection Current significant alcohol or drug abuse Inability to produce sputum samples of sufficient quality Subjects with a sputum neutrophil count greater than 10 million cells per ml Subjects who have taken an investigational drug within 3 months or 6 half-lives of the therapeutic intervention prior to Visit 1

Additional exclusion criteria for asthma patients:

Respiratory tract infection or asthma exacerbation in the 6 week period prior to Visit 1 (patients with mild to moderate asthma should be exacerbation free for a period of 12 months prior to Visit 1.

Patients with documented non-compliance to prescribed asthma controller therapy Treatment with biological agents (other than Xolair for severe asthma) within four months prior to Visit 1 Patients who have completed a pulmonary rehabilitation program in the six weeks prior to Visit 1 or who are currently in a pulmonary rehabilitation program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asthma and healthy subject
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- United Kingdom (4):
  - 352.2087.44001 Boehringer Ingelheim Investigational Site, Leicester
  - 352.2087.44004 Boehringer Ingelheim Investigational Site, London
  - 352.2087.44002 Boehringer Ingelheim Investigational Site, Manchester
  - 352.2087.44003 Boehringer Ingelheim Investigational Site, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a non-interventional, prospective, exploratory study. Asthma severity (mild, moderate or severe) was determined on the basis of medication use, spirometry (Forced Expiratory Volume in one second (FEV1) predicted values) and exacerbation history.
Groups:
- Healthy Volunteers: This group consisted of all healthy volunteers aged between 18 and 70 years without any significant comorbid condition.
- Mild Asthma: Patients with asthma are categorized as mild if they are taking Short-acting beta-agonist (SABA) or SABA/Short-acting muscarinic-antagonist (SAMA) per re nata (as required) (PRN), have no exacerbation in previous 12 months and have FEV1 ≥80 % of predicted.
- Moderate Asthma: Patients with asthma are categorized as moderate if they are taking at least low dose Inhaled corticosteroid (iCS) ± 2nd controller, have no exacerbation in previous 12 months and have FEV1 ≥ 60 - ≤ 85 % of predicted.
- Severe Asthma: Patients with asthma are categorized as severe if they are taking at least medium dose iCS ± 2nd controller and have at least 1 exacerbation (requiring treatment with systemic corticosteroids) in previous 12 months.
Period: Overall Study
Arm/Group | Healthy Volunteers | Mild Asthma | Moderate Asthma | Severe Asthma
Started | 10 | 12 | 20 | 27
Completed | 10 | 12 | 18 | 25
Not Completed | 0 | 0 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Observed Subjects Set (OBS): All subjects enrolled in the trial, following the receipt of informed consent, who are eligible to enter the observation period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Mild Asthma | Moderate Asthma | Severe Asthma | Total
Number analyzed (Participants) | 10 | 12 | 20 | 27 | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (14.6) | 36.1 (13.5) | 44.9 (12.6) | 50.2 (13.6) | 44.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 8 | 16 | 34
  Male | 6 | 6 | 12 | 11 | 35

OUTCOME MEASURES:

1. Primary Outcome: Level of Tumour Necrosis Factor-alpha (TNF-α) in Blood at Baseline (Visit 1)
Description: Level of Tumour Necrosis Factor-alpha (TNF-α) [picograms per milliliter (pg/mL)] in blood at baseline (Visit 1) is presented.
Time Frame: Baseline (Visit 1)
Population: Biomarker Subjects Set (BM) - All subjects, from the OBS [subjects enrolled in the trial, following the receipt of informed consent, and are eligible to enter the observation period], with at least one valid biomarker measurement either from blood or sputum at either visit.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Healthy Volunteers | Mild Asthma | Moderate Asthma | Severe Asthma
Number analyzed (Participants) | 8 | 10 | 13 | 25
pg/mL | 5.3 (5.1) | 9.3 (23.4) | 10.6 (13.1) | 15.7 (70.2)

2. Primary Outcome: Level of Interleukin-6 (IL-6) in Blood at Baseline (Visit 1)
Description: Level of Interleukin-6 (IL-6) (pg/mL) in blood at baseline (Visit 1) is presented.
Time Frame: Baseline (Visit 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Healthy Volunteers | Mild Asthma | Moderate Asthma | Severe Asthma
Number analyzed (Participants) | 8 | 10 | 13 | 25
pg/mL | 71.3 (109.0) | 65.2 (88.2) | 245.0 (426.3) | 133.9 (639.5)

3. Secondary Outcome: Level of Tumour Necrosis Factor-alpha (TNF-α) in Blood at Follow-up Visit 28 Days After Baseline (Visit 2)
Description: Level of Tumour Necrosis Factor-alpha (TNF-α) (pg/mL) in blood at follow-up visit 28 days after baseline (Visit 2) is presented.
Time Frame: follow-up visit 28 days after baseline (Visit 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Healthy Volunteers | Mild Asthma | Moderate Asthma | Severe Asthma
Number analyzed (Participants) | 10 | 12 | 16 | 25
pg/mL | 5.8 (9.6) | 8.1 (14.7) | 5.2 (5.5) | 16.4 (65.6)

4. Secondary Outcome: Level of Interleukin-6 (IL-6) in Blood at Follow-up Visit 28 Days After Baseline (Visit 2)
Description: Level of Interleukin-6 (IL-6) (pg/mL) in blood at follow-up visit 28 days after baseline (Visit 2) is presented.
Time Frame: follow-up visit 28 days after baseline (Visit 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Healthy Volunteers | Mild Asthma | Moderate Asthma | Severe Asthma
Number analyzed (Participants) | 10 | 12 | 16 | 25
pg/mL | 47.7 (59.7) | 86.1 (107.6) | 105.1 (94.1) | 37.4 (113.8)

ADVERSE EVENTS:
Time Frame: From baseline assessment (visit 1) till follow-up assessment (visit 2); up to 31 days
Description: Observed Subjects Set (OBS): All subjects enrolled in the trial, following the receipt of informed consent, who are eligible to enter the observation period.
Arm/Group | Healthy Volunteers | Mild Asthma | Moderate Asthma | Severe Asthma
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/20 | 0/27
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/20 | 0/27

LIMITATIONS AND CAVEATS:
The study is considered exploratory in nature as the definitive power needed to assess yet unknown endotypes cannot be prospectively specified. The study is, however, adequately designed as hypothesis generating study informing interventional studies

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.